CLINICAL TRIAL: NCT04008147
Title: The Effect of Oral Iron Supplements on Hepcidin, Insulin and Glucose Metabolism in Pregnancy
Brief Title: Hepcidin and Glucose Metabolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Principal Investigator, Isabelle Herter-Aeberli, PhD, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INDIA
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Iron Deficiency Anemia of Pregnancy; Iron Metabolism Disorders; Glucose Intolerance; Gestational Diabetes
MeSH Terms: conditions — Iron Metabolism Disorders; Glucose Intolerance; Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Iron Group (Active Comparator): 15 women taking 100 mg iron twice daily for 4 days (800 mg).
  Interventions: Dietary Supplement: 100mg iron fumarate
- Low Iron Group (Active Comparator): 15 women taking 30 mg iron once daily for 14 days (420 mg).
  Interventions: Dietary Supplement: Burgerstein Schwangerschaft & Stillzeit

INTERVENTIONS:
Dietary Supplement: 100mg iron fumarate — 100mg iron fumarate b.i.d. for 4 consecutive days
  Arms: High Iron Group
Dietary Supplement: Burgerstein Schwangerschaft & Stillzeit — contains 30 mg iron fumarate, given on 14 consecutive days
  Arms: Low Iron Group

SUMMARY:
Gestational diabetes mellitus (GDM), defined as hyperglycemia with blood glucose values above normal but below those diagnostic of DM, and iron deficiency (ID) with or without anemia (IDA) are common during pregnancy. Both disease patterns are associated with an increased risk of complications during pregnancy and at delivery and may have a variety of negative effects on different aspects of child development. Thus, GDM and ID/IDA during pregnancy should be prevented.

Whether iron supplementation with high oral doses acutely increases hepcidin during pregnancy, and whether this acute iron-induced increase in hepcidin decreases insulin sensitivity, is uncertain.

ELIGIBILITY:
Inclusion Criteria:

* week of pregnancy 24-28
* pre-pregnancy BMI <27.5kg/m2
* singleton pregnancy
* Hb > 8.0 g/dl

Willing to either:

* not take any iron supplements for 14 days (however, participants will receive a similar amount of total iron during the 4 study days that they would normally receive over 14 days) OR
* to take the multivitamin "Burgerstein Schwangerschaft and Stillzeit" supplements over the 14 days (contains 30 mg iron)

Exclusion Criteria:

* iron infusion within the past 6 months
* severely anemic Hb<8.0g/dl
* acute or chronic disease
* long-term medication
* medical problems known to affect iron homeostasis
* smoking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 30 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum hepcidin | before OGTT, 1 day before high/low iron supplementation
Serum hepcidin | after OGTT, 1 day before high/low iron supplementation
Serum hepcidin | before OGTT, after high/low iron supplementation at day 7
Serum hepcidin | after OGTT, after high/low iron supplementation at day 7
Serum iron | before OGTT, 1 day before high/low iron supplementation
Serum iron | after OGTT, 1 day before high/low iron supplementation
Serum iron | before OGTT, after high/low iron supplementation at day 7
Serum iron | after OGTT, after high/low iron supplementation at day 7
glucose | before OGTT, 1 day before high/low iron supplementation
glucose | after OGTT, 1 day before high/low iron supplementation
glucose | before OGTT, after high/low iron supplementation at day 7
glucose | after OGTT, after high/low iron supplementation at day 7
insulin | before OGTT, 1 day before high/low iron supplementation
insulin | after OGTT, 1 day before high/low iron supplementation
insulin | before OGTT, after high/low iron supplementation at day 7
insulin | after OGTT, after high/low iron supplementation at day 7
Serum hepcidin | At day 14, 7 days after high iron supplementation and 1 day after low iron supplementation
Serum iron | At day 14, 7 days after high iron supplementation and 1 day after low iron supplementation
glucose | At day 14, 7 days after high iron supplementation and 1 day after low iron supplementation
insulin | At day 14, 7 days after high iron supplementation and 1 day after low iron supplementation

SECONDARY OUTCOMES:
Serum ferritin | before OGTT, 1 day before high/low iron supplementation
Serum ferritin | after OGTT, 1 day before high/low iron supplementation
Serum ferritin | before OGTT, after high/low iron supplementation at day 7
Serum ferritin | after OGTT, after high/low iron supplementation at day 7
soluble transferrin receptor | before OGTT, 1 day before high/low iron supplementation
soluble transferrin receptor | after OGTT, 1 day before high/low iron supplementation
soluble transferrin receptor | before OGTT, after high/low iron supplementation at day 7
soluble transferrin receptor | after OGTT, after high/low iron supplementation at day 7
c-reactive protein | before OGTT, 1 day before high/low iron supplementation
c-reactive protein | after OGTT, 1 day before high/low iron supplementation
c-reactive protein | before OGTT, after high/low iron supplementation at day 7
c-reactive protein | after OGTT, after high/low iron supplementation at day 7
alpha glycoprotein | before OGTT, 1 day before high/low iron supplementation
alpha glycoprotein | after OGTT, 1 day before high/low iron supplementation
alpha glycoprotein | before OGTT, after high/low iron supplementation at day 7
alpha glycoprotein | after OGTT, after high/low iron supplementation at day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No